CLINICAL TRIAL: NCT02066727
Title: Effects of Dexmedetomidine as an Adjuvant on the Median Effective Concentration of Lidocaine for Obturator Nerve Block - A Perspective, Randomized，Blind Study
Brief Title: Lidocaine Combined Dexmedetomidine for Obturator Nerve Block
Acronym: ONB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guolin Wang (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor-Investigator, Guolin Wang, Tianjin Medical University General Hospital, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GW002
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Nerve Block
Keywords: Dexmedetomidine; obturator nerve block; lidocaine; EC50
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine is administrated as an adjuvant of lidocaine at a dose of 1.0 μg/ kg.
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Placebo Comparator): Normal Saline is administrated as an adjuvant of lidocaine.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is administrated as an adjuvant of lidocaine at a dose of 1.0 μg/ kg.
  Arms: Dexmedetomidine
Drug: Normal Saline — Normal Saline is administrated as an adjuvant of lidocaine.
  Arms: Normal Saline

SUMMARY:
Hypothesis: Dexmedetomidine as an adjuvant of lidocaine can decrease the median effective concentration(EC50) of lidocaine for obturator nerve block during transurethral resection of bladder tumor

DETAILED DESCRIPTION:
A selective obturator nerve block(ONB) is an effective alternative to suppress the obturator nerve reflex which is defined as a sudden, violent adductor muscle spasm when the obturator nerve is stimulated directly by the electronic resector during transurethral resection of the tumor on the lateral bladder wall. Studies showed Dexmedetomidine as an adjuvant to local anesthetic prolongs peripheral nerve block duration without any nerve toxicity. In the following randomized, non-crossover study, the investigators test if Dexmedetomidine as an adjuvant can decrease the median effective concentration(EC50) of lidocaine for obturator nerve block during transurethral resection of bladder tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to undergo elective operation of TURBT on lateral wall for whom ONB was needed diagnosed through cystoscopy or CT examination preoperatively.
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of abnormal coagulation function.
2. Subject has a diagnosis of Diabetes mellitus.
3. Subject has a preexisting neurologic deficits of the lower extremities.
4. Subject has a history of alcohol or drug abuse.
5. Subject is pregnant or breast-feeding.
6. Subject is obese (body mass index >30kg/m2).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD.PHD, Study Director — Tainjin Medical University General Hospita
Locations (1):
- Tainjin Medical University General Hospita& the Second Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Lu Y, Sun J, Zhuang X, Lv G, Li Y, Wang H, Wang G. Perineural Dexmedetomidine as an Adjuvant Reduces the Median Effective Concentration of Lidocaine for Obturator Nerve Blocking: A Double-Blinded Randomized Controlled Trial. PLoS One. 2016 Jun 24;11(6):e0158226. doi: 10.1371/journal.pone.0158226. eCollection 2016. PMID 27341450

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The patients with the following condition was excluded from the study: ASA III orIV; weight <50 or >100 kg；BMI<19 or >30kg/m2；age younger than 18 yr or older than 80yr；preexisting neurologic deficits of the lower extremities, DM; alcohol or drug abuse; abnormal coagulation function
Period: Overall Study
Arm/Group | Normal Saline | Dexmedetomidine
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Dexmedetomidine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 68 (9) | 65 (12)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 39
  >=65 years | 12 | 9 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Median Effective Concentration(EC50)
Description: Median effective concentration(EC50) was not calculated per-participants, the "up-and-down" sequential allocation method was used to determine the median effective concentration(EC50) of lidocaine, running the two groups in parallel. The concentration of lidocaine for the second and subsequent patients in each group were dictated by the response of the previous patient in the group, such that an effective block led to a decreased concentration of the next patient, an ineffective block led to an increased concentration.
  For each group, we collected: the logarithm of lidocaine concentration, the number of effective block, ineffective block, total number of the patient, and successful rate. Then lgEC50 and slgEC50 was calculated as formulas. The logarithm of confidence intervals(95% CI) was calculated as lgEC50±1.96slgEC50. All of the calculation can be performed by SPSS19.0 for windows.
Time Frame: 10min
Measure: Number (95% Confidence Interval); unit: mg/ml(the concentration of lidocaine)
Arm/Group | Normal Saline | Dexmedetomidine
Number analyzed (Participants) | 30 | 30
mg/ml(the concentration of lidocaine) | 5.7 [5.4 to 6.2] | 2.9 [2.8 to 3.8]

2. Secondary Outcome: Complication Related With Nerve Block
Description: Complication related with nerve block is defined as the presence of either bradycardia, delayed recovery, persistent groin pain, neuropathy during operation and postoperatively
Time Frame: during operation, 0.5,24hour postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Form the completion of obturator nerve block to 24 hours after operation.
Arm/Group | Normal Saline | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes